CLINICAL TRIAL: NCT02940392
Title: Rezum First in Man Feasibility Study for the Treatment of BPH With the Rezum System
Brief Title: Rezum FIM Optimization Study
Acronym: Rezum FIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1633-001
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-02

CONDITIONS: Benign Prostatic Hyperplasia; Adenoma, Prostatic; Prostatic Adenoma; Prostatic Hyperplasia, Benign; Prostatic Hypertrophy; Prostatic Hypertrophy, Benign; Rezum
Keywords: Rezum
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rezum Treatment (Experimental): Patients will receive the Rezūm transurethral needle ablation procedure to treat benign prostatic hyperplasia.
  Interventions: Device: Rezum System

INTERVENTIONS:
Device: Rezum System — The Rezūm System is designed to treat patients with bothersome urinary symptoms associated with benign prostatic hyperplasia (BPH). The Rezūm System utilizes radiofrequency current to generate "wet" thermal energy in the form of water vapor, which is then injected into the transition zone and/or median lobe of the prostate tissue in controlled 9-second doses. The vapor that is injected into the prostate tissue rapidly disperses through the interstitial space between the tissue cells. As the vapor cools, it condenses immediately on contact with tissue and the stored thermal energy is released, denaturing the cell membranes and causing cell death.
  The denatured cells are absorbed by the body, which reduces the volume of prostate tissue adjacent to the urethra. The vapor condensation process also causes a rapid collapse of vasculature in the treatment zone, resulting in a bloodless procedure.
  Other Names: Rezum Procedure; Rezum; Water Vapor Ablation; Rezum Delivery Device; Rezum Generator

SUMMARY:
Evaluate the effect of the NxThera BPH Rezum System on prostate tissue in subjects suffering from LUTS symptoms secondary to benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
Subjects with BPH symptoms were treated with the Rezum device with a range of thermal energies (as measured by calorie output) to optimize the setting for maximum lesion size with minimal intra and post-procedure discomfort. Lesion size and ablated tissue resorption rate was followed post-procedure at 1 week, 1 month, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects > 45 years of age who have symptomatic / obstructive symptoms secondary to BPH requiring invasive intervention.
2. IPSS score of ≥ 15.
3. Qmax: Peak flow rate ≤ 15 ml/sec.
4. Post-void residual (PVR) < 300 ml.
5. Prostate transverse diameter > 30 mm.
6. Prostate volume between 20 to 120 gm.
7. Voided volume ≥ 125 ml.
8. Subject able to complete the study protocol in the opinion of the Principal Investigator.
9. Subject must be willing to undergo the procedure without anesthesia.

Exclusion Criteria:

1. History of any illness or surgery that in the opinion of the Principal Investigator may confound the results of the study.
2. Presence of a penile implant.
3. Any prior minimally invasive intervention (e.g. TUNA,Laser, Microwave) or surgical intervention for the symptoms of BPH.
4. Currently enrolled in another clinical trial.
5. Confirmed or suspected malignancy of prostate or bladder.
6. Previous rectal surgery (other than hemorrhoidectomy) or history of rectal disease.
7. Previous pelvic irradiation or radical pelvic surgery.
8. Documented active urinary tract infection by culture or bacterial prostatitis within last year documented by culture (UTI is defined as >100,000 colonies per ml urine from midstream clean catch or catheterization specimen).
9. Neurogenic bladder or sphincter abnormalities.
10. Urethral strictures, bladder neck contracture or muscle spasms.
11. Bleeding disorder (note that use of anti-platelet medication is not an exclusion criterion).
12. Subjects who are interested in maintaining fertility.
13. Use of concomitant (or recent) medications to include the following:

    1. Beta blockers, antihistamines, anticonvulsants, and antispasmodics within 1 week of treatment, unless there is documented evidence of stable dosing for last 6 months (e.g., no dose changes).
    2. Alpha blockers, antidepressants, anticholinergics, androgens, or gonadotropin-releasing hormonal analogs within 2 weeks of treatment.
    3. 5-alpha reductase inhibitor within the last 6 months
14. Subject is unable or unwilling to go through a "washout" period for the above medications prior to treatment.
15. Subject has chronic urinary retention.
16. Significant urge incontinence.
17. Poor detrusor muscle function.
18. Neurological disorders which might affect bladder or sphincter function.
19. Bladder stones.
20. Renal impairment.
21. In the opinion of the Principal Investigator, subject will not be able to adequately tolerate a rigid cystoscopy-type procedure.
22. Unable or unwilling to sign the Informed Consent Form (ICF) and/or comply with all the required follow-up requirements.
23. Any cognitive disorder that interferes with or precludes a subject from directly and accurately communicating with the Principal Investigator regarding the study.
24. Peripheral arterial disease with intermittent claudication or Leriches Syndrome (i.e., claudication of the buttocks or perineum).
25. Biopsy of the prostate within 30 days prior to the Rezūm procedure.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-03-19 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Canela, La Romana, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single arm, single center interventional study recruited subjects who met inclusion/exclusion criteria and consented to participate. Subjects on BPH medication underwent a washout period prior to treatment. Subjects who successfully completed the washout period and still met the inclusion/exclusion criteria were enrolled in the study. Subjects were considered officially enrolled only if treatment with the NxThera Rezūm System was attempted.
Groups:
- Rezum Treatment: Participants underwent the Rezūm transurethral needle ablation procedure to treat benign prostatic hyperplasia. They were followed for 5 years for adverse events and quality of life data.
  Rezum System: The Rezūm System is designed to treat patients with bothersome urinary symptoms associated with benign prostatic hyperplasia (BPH). The Rezūm System utilizes radiofrequency current to generate "wet" thermal energy in the form of water vapor, which is then injected into the transition zone and/or median lobe of the prostate tissue in controlled 9-second doses. The vapor that is injected into the prostate tissue rapidly disperses through the interstitial space between the tissue cells. As the vapor cools, it condenses immediately on contact with tissue and the stored thermal energy is released, denaturing the cell membranes and causing cell death.
  The denatured cells are absorbed by the body, which reduces the volume of prostate tissue adjacent to the urethra. The vapor condensation process also causes a rapid collapse of vasculature in the treatment zone, resulting in a bloodless procedure.
Period: Overall Study
Arm/Group | Rezum Treatment
Started | 15
Completed | 7
Not Completed | 8
Not completed — Lost to Follow-up | 3
Not completed — Retreatment | 3
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic/Latino | 14
  Race/Ethnicity: Caucasian | 1
Region of Enrollment [Number; unit: participants]
  Dominican Republic | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in International Prostate Symptom Score
Description: International Prostate Symptom Score (IPSS) scores were recorded at Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, then annually to 5 years. The mean change in IPSS was calculated.
  The IPSS is a validated questionnaire used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of benign prostatic hyperplasia (BPH). Scoring ranges from 0 to 35 with overall scores of 0-7 correlated to mildly symptomatic, 8-19 correlated to moderately symptomatic and 20-35 correlated to severely symptomatic. A reduction in score from baseline corresponds to improved outcome post procedure.
Time Frame: Baseline to 1 week, 1 month, 3 months, 6 months, 1 year, annually to 5 years
Population: Mean change in score was calculated for the number of subjects providing data at each follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 15
score on a scale
  IPSS Change at 1 Week | -6.1 (13.8)
  IPSS Change at 1 Month | -12.9 (12.8)
  IPSS change at 3 months: number analyzed (Participants) | 14
  IPSS change at 3 months | -14.6 (9.1)
  IPSS change at 6 months: number analyzed (Participants) | 14
  IPSS change at 6 months | -14.8 (11.0)
  IPSS change at 12 months: number analyzed (Participants) | 13
  IPSS change at 12 months | -13.6 (7.5)
  IPSS change at 24 months: number analyzed (Participants) | 8
  IPSS change at 24 months | -13.9 (5.1)
  IPSS change at 36 months: number analyzed (Participants) | 9
  IPSS change at 36 months | -7.6 (6.4)
  IPSS change at 48 months: number analyzed (Participants) | 6
  IPSS change at 48 months | -13.0 (7.4)
  IPSS change at 60 months: number analyzed (Participants) | 7
  IPSS change at 60 months | -7.6 (6.3)

2. Other Pre Specified Outcome: Intra-procedural and Post-procedural Pain
Description: Intra-procedural and post-procedural pain for each subject was assessed using the Wong Baker Pain Rating scale (0-10 with 0 indicating no pain and 10 indicating worst pain imaginable). Each subject selected the response on the pain scale that he felt best represented his pain level. Unless otherwise noted, the subjects were not given pain medications or anesthesia. All subjects were given an anti-anxiety medication plus a Non-Steroidal Anti-Inflammatory Drug (NSAID) pre-procedure.
Time Frame: Procedure Day, 1 day post procedure, 1 week post procedure, 1 month post procedure, 3 months post procedure ,6 months post procedure
Population: Pain score was not collected for 1 subject at each of the following visits: 1 day, 3 month, and 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 15
score on a scale
  average pain score post-procedure (day of procedure) | 3.5 (2.7)
  average pain 1 day post-procedure: number analyzed (Participants) | 14
  average pain 1 day post-procedure | 0.1 (0.3)
  average pain 1 week post-procedure | 0.2 (0.6)
  average pain 1 month post-procedure | 0.5 (2.1)
  average pain 3 months post-procedure: number analyzed (Participants) | 14
  average pain 3 months post-procedure | 0.0 (0.0)
  average pain 6 months post-procedure: number analyzed (Participants) | 14
  average pain 6 months post-procedure | 0.0 (0.0)

3. Other Pre Specified Outcome: Number of Subjects Requiring Catheterization Post Procedure
Description: All subjects were kept at the clinic for observation for 24 hours post-procedure. The number of subjects requiring post-procedure catheterization were recorded.
Time Frame: 1 day post procedure, 1 week post procedure, 1 month post procedure
Population: Number of subjects requiring post-procedure catheterization. Two (2) subjects were catheterized prior to the Rezūm study enrollment and treatment. The decision was made to move forward with treating both subjects. All subjects were observed for 24 hours in the clinic post-procedure. Post-procedure catheterization was allowed if determined that the subject had symptoms of retention (defined as failure to void within 8 hours post procedure) or required catheterization for other safety reasons.
Measure: Number; unit: participants
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 15
participants
  Subjects catheterized at 1 day post procedure | 9
  Subjects catheterized at 1 week post procedure | 8
  Subjects catheterized at 1 month post procedure | 3

4. Other Pre Specified Outcome: Post Procedure Catheterization Duration
Description: Measures the duration (days) of catheterization for subjects who required catheterization post procedure. Post-procedure catheterization was allowed if the Principal Investigator determined that the subject had symptoms of retention (defined as failure to void within 8 hours post procedure) or required catheterization for other safety reasons.
Time Frame: 1 month post procedure
Population: Data provided for subjects who underwent the Rezūm ablation procedure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 15
days
  Overall catheterization duration (days) per subject: number analyzed (Participants) | 10
  Overall catheterization duration (days) per subject | 7.6 (10.9)
  Overall catheterization duration (days) per episode (13 episodes in 10 subjects): number analyzed (Participants) | 10
  Overall catheterization duration (days) per episode (13 episodes in 10 subjects) | 5.8 (6.8)

5. Other Pre Specified Outcome: Lesion Characteristics Via MRI (Changes in Lesion Volume)
Description: Lesion size and treated tissue resorption rate was measured by gadolinium enhanced MRI on all subjects at 1 week, 1 month, 3 months, and 6 months post-procedure. The percent change in lesion volume was calculated.
Time Frame: 1 week , 1 month, 3 months, 6 months post procedure
Population: One subject (each) did not have MRI available at the 3 month and 6 month follow-up visit.
Measure: Mean (Standard Deviation); unit: percentage of change in lesion volume
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 15
percentage of change in lesion volume
  Mean percent change from 1 week to 1 month | -53.7 (17.8)
  Mean percent change from 1 week to 3 months: number analyzed (Participants) | 14
  Mean percent change from 1 week to 3 months | -88.9 (8.1)
  Mean percent change from 1 week to 6 months: number analyzed (Participants) | 14
  Mean percent change from 1 week to 6 months | -95.8 (4.8)

6. Other Pre Specified Outcome: Lesion Characteristics Via MRI (Changes in Prostate Volume)
Description: Lesion size and treated tissue resorption rate was measured by gadolinium enhanced MRI on all subjects at 1 week, 1 month, 3 months, and 6 months post-procedure. The percent change in prostate volume was calculated.
Time Frame: 1 week, 1 month, 3 months, 6 months post-procedure
Population: One subject (each) did not have MRI data available at the 3 month and 6 month visit
Measure: Mean (Standard Deviation); unit: percentage of change in prostate volume
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 15
percentage of change in prostate volume
  Mean percent change from 1 week to 1 month | -14.7 (13.2)
  Mean percent change from 1 week to 3 months: number analyzed (Participants) | 14
  Mean percent change from 1 week to 3 months | -25.6 (11.4)
  Mean percent change from 1 week to 6 months: number analyzed (Participants) | 14
  Mean percent change from 1 week to 6 months | -32.3 (10.8)

7. Other Pre Specified Outcome: Lesion Characteristics Via MRI (Changes in Transition Zone Volume)
Description: Lesion size and treated tissue resorption rate was measured by gadolinium enhanced MRI on all subjects at 1 week, 1 month, 3 months, and 6 months post-procedure. The percent change in transition (TZ) zone volume was calculated
Time Frame: 1 week, 1 month, 3 months, 6 months post-procedure
Population: One subject (each) did not have MRI available at the 3 month and 6 month visit
Measure: Mean (Standard Deviation); unit: percentage of change in TZ volume
Arm/Group | Rezum Treatment
Number analyzed (Participants) | 15
percentage of change in TZ volume
  Mean percent change from 1 week to 1 month | -18.6 (15.0)
  Mean percent change from 1 week to 3 months: number analyzed (Participants) | 14
  Mean percent change from 1 week to 3 months | -30.4 (13.6)
  Mean percent change from 1 week to 6 months: number analyzed (Participants) | 14
  Mean percent change from 1 week to 6 months | -37.7 (14.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of index procedure through the 60 month follow-up assessment.
Description: AEs were adjudicated by an independent urologist who served on the Rezūm II Pivotal Study Clinical Events Committee (CEC).
  51 adverse events were reported by 14 subjects. Of the 51 events, 25 events (49.0%) were adjudicated as device related and 32 (62.7%) as procedure related.
Arm/Group | Rezum Treatment
All-Cause Mortality (participants affected / at risk) | 2/15
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rezum Treatment (N=15)
Subject was surgically treated for a pre-existing hernia. (Renal and urinary disorders) | 1 (1) — This condition was present prior to treatment. Details were not available; the procedure was done at another site.
Adenocarcinoma (Renal and urinary disorders) | 1 (1) — At 1 year follow up subjects PSA was 15.4. A prostate biopsy was scheduled. Biopsy results positive for Adenocarcinoma. Subject had a prostatectomy and was exited from the study.
Urinary Retention (Renal and urinary disorders) | 1 (1) — Subject reported urinary retention at 3 month visit; treated medically. Subject reported continued urinary retention with fever and dysuria. A UTI was diagnosed; treated medically. Subsequently treated for retention followed by Prostatectomy.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rezum Treatment (N=15)
Urinary Tract Infection (UTI) - Suspected (Renal and urinary disorders) | 7 (9)
Urinary Retention (Renal and urinary disorders) | 6 (6)
Dysuria (Renal and urinary disorders) | 4 (5)
Hematuria (Renal and urinary disorders) | 5 (5)
Fever (General disorders) | 3 (4)
Poor Stream (Renal and urinary disorders) | 3 (4)
Urinary Urgency (Renal and urinary disorders) | 2 (3)
Infection (non UTI) (Infections and infestations) | 2 (2)
Other (General disorders) | 1 (1)
Terminal Dribbling (Renal and urinary disorders) | 2 (2)
Urinary Frequency (Renal and urinary disorders) | 2 (2)
Hematuria with Clots and Retention (Renal and urinary disorders) | 1 (1)
Prostatic Urethral Injury (Renal and urinary disorders) | 1 (1)
UTI - Prophylaxis (Renal and urinary disorders) | 1 (1)
Ureteral Calculi (Renal and urinary disorders) | 1 (1)
Urinary Incontinence - Urge (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT02940392/Prot_SAP_000.pdf